CLINICAL TRIAL: NCT03433430
Title: This is an Exploratory Multi-center, Pilot Study to Evaluate the Safety, Efficacy and Ergonomics of Cutera truSculpt Device. Subjects May Receive up to Three Treatments and Will be Followed at 12 Weeks Post the First and Final Treatment.
Brief Title: Multi-Center Pilot Study of truSculpt Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-17-TS16
Record Dates: First submitted 2018-02-05; First posted 2018-02-14 (Actual); Results first posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Bulging; Body Fat

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- truSculpt (Other): truSculpt treatment
  Interventions: Device: truSculpt

INTERVENTIONS:
Device: truSculpt — Subjects will receive utreatments and will be followed at 12 weeks post final treatment.

SUMMARY:
An exploratory pilot study to evaluate the safety, efficacy and ergonomics of Cutera truSculpt device

DETAILED DESCRIPTION:
This is a multi-center, pilot study in approximately 40 subjects, ages 18 to 65. Subjects will receive treatments and will be followed at 12 weeks post final treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be able to read, understand and sign the Informed Consent Form.
2. Female or Male, 18 to 65 years of age (inclusive).
3. Subject has visible fat bulges in the area to be treated.
4. Non-smoking for at least 6 months and willing to refrain from smoking for the duration of the study.
5. Subject must agree to not undergo any other procedure(s) in the treatment region during the study period.
6. Subject must adhere to the follow-up schedule and study instructions.
7. Subject must adhere to the same diet and/or exercise routine throughout the study, and agree to maintain the same weight throughout the study.
8. Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation, (educational and/or marketing), publications, and any additional marketing purposes.
9. For female subjects: not pregnant or lactating and is either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study.

Exclusion Criteria:

1. Participation in a clinical trial of another device or drug within 3 months of study participation, or during the study period.
2. Any type of prior cosmetic treatment to the target area within 6 months of study participation.
3. Any prior invasive cosmetic surgery to the target area, such as liposuction.
4. Has a pacemaker, internal defibrillator, implantable cardioverter-defibrillator, nerve stimulator implant, cochlear implant or any other electronically, magnetically or mechanically activated implant.
5. Has metal implant(s) within the body, such as artificial heart valves.
6. Significant uncontrolled concurrent illness that in the opinion of the Investigator would make the subject unsuitable for inclusion.
7. History of any disease or condition that could impair wound healing.
8. History of keloid formation, hypertrophic scarring or abnormal/delayed wound healing.
9. Skin abnormality in the treatment area that in the opinion of the Investigator would make the subject unsuitable for inclusion.
10. Currently undergoing systemic chemotherapy or radiation treatment for cancer, or history of treatment in the target area within 3 months of study participation.
11. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study or a condition that would compromise the subject's ability to comply with the study requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2018-03-07 (Actual); Study Completion 2018-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Ronan, MD, Principal Investigator — Cutera Research Center; Ashish Bhatia, MD, Principal Investigator — The Dermatology Institute of DuPage Medical Group; Joely Kaufman, MD, FAAD, Principal Investigator — Skin Associates of South Florida
Locations (3):
- United States (3):
  - Cutera Research Center, Brisbane, California
  - Skin Associates of South Florida, Coral Gables, Florida
  - The Dermatology Institute of DuPage Medical Group, Naperville, Illinois

RESULTS

PARTICIPANT FLOW:
Groups:
- truSculpt: Treatment with the truSculpt RF device
Period: Overall Study
Arm/Group | truSculpt
Started | 9
Completed | 8
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | truSculpt
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Body Fat Assessment by Investigator
Description: Degree of Improvement in body fat as assessed by Investigator using the Global Aesthetic Improvement Scale (GAIS:) +4=Very Significant Improvement, +3=Significant Improvement, +2=Moderate Improvement, +1=Mild Improvement, and 0=No Change Higher scores indicate better outcomes
Time Frame: 12 weeks post final treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | truSculpt
Number analyzed (Participants) | 8
score on a scale | 1.88 (1.13)

ADVERSE EVENTS:
Time Frame: 12 weeks post-final treatment, up to 6 months
Arm/Group | truSculpt
All-Cause Mortality (participants affected / at risk) | 0/9
Serious Adverse Events (participants affected / at risk) | 0/9
Other Adverse Events (participants affected / at risk) | 9/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | truSculpt (N=9)
Erythema (Skin and subcutaneous tissue disorders) | 9
Pain (Skin and subcutaneous tissue disorders) | 2
Tenderness (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-07-28): https://cdn.clinicaltrials.gov/large-docs/30/NCT03433430/Prot_001.pdf